CLINICAL TRIAL: NCT02651740
Title: Efficacy and Safety Evaluation of Rifaximin Combined Fecal Microbiota Transplantation in the Treatment of Irritable Bowel Syndrome With Predominant Diarrhea
Brief Title: Gut Microbiota Reconstruction in the Treatment of Irritable Bowel Syndrome With Predominant Diarrhea
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SXZ-WSD01-2015
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Rifaximin; Fecal microbiota transplantation; Gut microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combining therapy (Experimental): taking rifaximin for 3 days and then receiving fecal microbiota transplantation with donor stool through enteral nutrition tube
  Interventions: Drug: Rifaximin; Procedure: Fecal microbiota transplantation

INTERVENTIONS:
Drug: Rifaximin — 400mg tid* 3d
  Other Names: Brand name: XIFAXAN; Production company: SALIX PHARMS
Procedure: Fecal microbiota transplantation — Using filtered fresh donor stool, 100-200ml per time throuth enteral nutrition tube for at least one time

SUMMARY:
The purpose of this study is to evaluate the efficacy as well as safety of rifaximin combined fecal microbiota transplantation(Gut microbiota reconstruction) in the treatment of IBS-D.

DETAILED DESCRIPTION:
In this prospective study, there is only one group with no placebo/blank control. All qualified IBS-D patients could be admitted to hospital for at least one time of combing therapy (taking rifaximin for 3 days and then receiving fecal microbiota transplantation) and follow-up until 6 months after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65, no gender limitation;
* Had received a diagnosis of IBS-D (as assessed according to the Rome III diagnosis criteria of IBS) and had undergone a colonoscopic examination within the previous 2 years with no organic lesions observed;
* Has current symptoms of IBS-D: ①Abdominal pain (at least 2 days in a week with no limitation of severity); ②Stool consistency (rated the consistency of their stools of Bristol types 6/7 at least once a day and at least 2 days in a week);
* Can do follow-up at required time points and signed written informed consent before the study.

Exclusion Criteria:

* Allergic to rifaximin;
* Taking alosetron, tegaserod, lubiprostone, warfarin, or antipsychotic, antispasmodic, antidiarrheal, probiotic, or narcotic drugs within the previous 1 month;
* Had infective diarrhea history or had taken antibiotics within the previous 14 days;
* Patients with a history of inflammatory bowel disease ;
* Previous abdominal surgery (other than cholecystectomy or appendectomy);
* Human immunodeficiency virus infection or other immunodeficiency conditions such as congenital immunodeficiency or currently taking immune-suppression drugs;
* Unstable diabetes, hypertension, thyroid disease, etc;
* Accompanied malignant tumor or severe heart/lung/renal/hepatic/brain/blood diseases;
* Accompanied severe neural/psychotic diseases such as epilepsy, depression, mania, schizophrenia, etc;
* Other conditions that doctor thought not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with relief of IBS condition | 6 months after the treatment
  The "responder" should at the same time get relief of at least one item of abdominal discomfort related symptoms(including abdominal pain score(0-10 with 0 indicates no pain and 10 indicates very great deal of pain) and bloating/abdominal discomfort score(0-10 with 0 indicates no discomfort and 10 indicates very great deal of discomfort), both items' effectiveness are defined as decreasing at least 30% compared with baseline) and at least one item of defecation related abnomalities(including average daily defecation(effectiveness defined as decreasing at least 30% compared with baseline) and stool consistency(effectiveness defined as feces could reach at least Bristol type 5) ).

SECONDARY OUTCOMES:
Number of patients with relief of IBS related anxiety or depression status | 1 month/2 month/3 month/6 month after the treatment
  The number of patients who have at least 30% decreasing compared with baseline in the score of SAS/SDS/HADS rating scale
Number of patients with relief of IBS single symptoms | 2 week/1 month/2 month/3 month/6 month after the treatment
  The number of patients who have relief of IBS global score(0-10 with 0 indicates no discomfort and 10 indicates very great deal of discomfort), pain score(0-10 with 0 indicates no pain and 10 indicates very great deal of pain), bloating/abdominal discomfort score(0-10 with 0 indicates no discomfort and 10 indicateds very great deal of discomfort), urgency score(0-3 with 0 indicates no urgency and 3 indicates great deal of urgency), average daily defecation, stool consistency(according to Bristol criteria). Except stool consistency, other items' effectiveness are defined as decreasing at least 30% compared with baseline during the whole period of follow-up. Stool consistency's effectiveness is defined as feces could reach at least Bristol type 5 during the whole period of follow-up.

OTHER OUTCOMES:
The rate and type of adverse effects | The day before check-out and 2 week/1 month/2 month/3 month/6 month after the treatment
  It means any events that occur in the trial process related or unrelated to the drug/fecal microbiota transplantation that do harm to the patients' health, including symptoms/physical signs/abnormal lab values

CONTACTS AND LOCATIONS:
Overall Officials: Xizhong Shen, PhD, Study Chair — Zhongshan Hospital, Shanghai, China
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided